CLINICAL TRIAL: NCT02346357
Title: Ultrasound-Guided Obturator Nerve Block for Ambulatory Hip Arthroscopy: A Prospective, Randomized Controlled Trial
Brief Title: Ultrasound-Guided Obturator Nerve Block for Ambulatory Hip Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benaroya Research Institute (Other)
Responsible Party: Principal Investigator, Francis V. Salinas , MD, Anesthesiologist, Benaroya Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB14003
Record Dates: First submitted 2014-11-20; First posted 2015-01-27 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Pain
Keywords: hip arthroscopy; analgesia
MeSH Terms: conditions — Pain; Agnosia | interventions — Nerve Block; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Obturator nerve block (Active Comparator): Ultrasound-guided single-injection obturator nerve block with 20 mL ropivacaine 0.5%
  Interventions: Procedure: Obturator Nerve Block; Drug: Ropivacaine
- Sham block (Placebo Comparator): Placebo arm. Ultrasound-guided injection of 3-5 mL normal saline in the subcutaneous tissue in the same location as would for an obturator nerve block.
  Interventions: Procedure: Obturator Nerve Block; Drug: Placebo Saline

INTERVENTIONS:
Procedure: Obturator Nerve Block — Ultrasound-guided obturator nerve block with 20 mL of treatment drug (Ropivacaine 0.5% [local anesthetic]) 30 minutes prior to induction of anesthesia.
  Other Names: Nerve block
Drug: Ropivacaine
  Arms: Obturator nerve block
Drug: Placebo Saline
  Arms: Sham block

SUMMARY:
Hip arthroscopy is commonly associated with moderate-to-severe postoperative pain. The purpose of this study is to investigate the analgesic efficacy of preoperative obturator nerve block as measured by postoperative pain scores and postoperative analgesic requirements. The primary outcome will be the patient's first reported pain scores in the post anesthesia care unit (PACU).

DETAILED DESCRIPTION:
RESEARCH DESIGN AND METHODS Patient selection The proposed study will be a prospective randomized placebo-controlled trial. Eligibility criteria will include patients having primary unilateral ambulatory hip arthroscopy for femoral acetabular impingement, age 18 to 65 years, ASA physical status I to III, and ability to follow the protocol.

Exclusion criteria: patient refusal, inability to comprehend the consent form, age < 18, and > 65 years of age; contraindications to obturator nerve blockade (pre-existing neuromuscular or peripheral nerve disorder, localized infection, or bleeding disorder); allergy to opioids or local anesthetics; allergy to celecoxib or sulfa medications or nonsteroidal anti-inflammatory medications (NSAIDs); chronic opioid use (> 1 month of 60 mg morphine PO equivalents daily); and, women who are pregnant or breastfeeding.

Consent Patients will be enrolled preoperatively in either the orthopedic surgery clinic or through the anesthesia preoperative clinic after the hip arthroscopy surgery is scheduled

Randomization, Blinding, and Allocation

Study medications will be administered by the primary investigator who will perform or closely supervise all ultrasound-guided obturator nerve blocks. Randomization will be performed with use of computerized random number generator and then each assignment will be placed into an opaque sealed envelope. Upon enrollment into the study and consent obtained, the next sealed envelope (numbered sequentially) will be opened and the patient allocated to either:

* Group 1 (Treatment), Ultrasound-guided obturator nerve block: 20 ml ropivacaine 0.5%
* Group 2 (Placebo), Ultrasound-guided saline placebo block: 5 mL sterile saline 0.9% The primary investigator will not be involved in any subsequent postoperative data collection. The sub-investigators will perform all subsequent data collection and will be blinded to group allocation.

Intervention Following randomization, the principle investigator will perform the block procedure 30 minutes prior to expected transfer back to the operating room.

Anesthetic care All intraoperative anesthetic care will be standardized as well, including general endotracheal anesthesia induction using propofol 1.5-2mg/kg IV, succinylcholine 1-1.5mg/kg IV or rocuronium 0.6-1mg/kg IV (based on the clinical discretion of the blinded anesthesia provider). In order to provide adequate intraoperative analgesia for both groups for the expected duration of the procedure, 1 mg of intravenous hydromorphone will be administered 10 minutes prior to surgical incision.

No further intraoperative opioids will be administered. Neuromuscular blockade will be maintained with rocuronium as indicated by surgical requirements and titrated by neuromuscular monitoring, and reversed in standard fashion prior to emergence from general anesthesia. At the end of the procedure, the surgeon will inject ropivacaine 0.25% 30 mL in each of the 2 arthroscopic portal sites for a total of 60 ml ropivacaine 0.25% in all subjects as is standard practice for all hip arthroscopy patients.

Subjects will be given a log to record their postoperative pain scores and oxycodone consumption for the 1st 24 hours after discharge.

Outcomes The primary outcome will be the pain immediately upon arrival to the post anesthesia care unit. This will be measured by an 11-point numerical rating scale (NRS 0 = no pain, and 10 = worst pain imaginable).

Secondary outcomes will include NRS pain scores at additional time frames for pain score self-assessments will include:

1. 3-4 hours after arriving home
2. Within 1 hour prior to going to sleep
3. Within 1 hour after waking up the following day.
4. 24 hours after surgery

Additional secondary outcomes will also include: cumulative 24-hour postoperative opioid consumption, percentage of patients with postoperative nausea and vomiting, sleep disturbance (difficulty going to sleep or waking up from sleep due to postoperative pain).

Expected Time Frame

Typically, 4-5 hip arthroscopies per week are performed. Thus the expected timetable for recruitment will take at least 6-12 months

ELIGIBILITY:
Inclusion Criteria:

* Primary unilateral ambulatory hip arthroscopy
* Age 18 to 65 years
* ASA physical status I to III
* Ability to follow the protocol.

Exclusion Criteria:

* Age <18 or >65 years of age
* Contraindications to peripheral nerve blockade
* Allergy to opioids or local anesthetics
* Allergy to sulfa medications or nonsteroidal anti-inflammatory medications
* Chronic opioid
* Patient refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Immediate pain score upon arrival to phase 1 PACU (NRS pain score) | Within 5-30 minutes upon leaving operating room and arrival to Phase I recovery
  Initial NRS pain score upon arrival in the post anesthesia cafe unit (PACU)

SECONDARY OUTCOMES:
Post anesthesia care unit discharge (Time required to meet discharge criteria from phase 2 PACU) | Wihtin 6 hours from end of surgery.
  Time required to meet discharge criteria from phase 2 PACU, able to be discharged home
Nausea (Number of episodes of nausea and vomiting during the 1st 24 hours postoperatively) | 1st 24 hours after surgery
  Number of episodes of nausea and vomiting during the 1st 24 hours postoperatively
Sleep quality on on the day of surgery (Did subjects have difficulty going to sleep or wake up from sleep due to pain?) | Within 12-24 hours after discharge to home (from the hospital); typically the same night of the day of surgery.
  Did subjects have difficulty going to sleep or wake up from sleep due to pain?
Opioid (analgesic) consumption | From the start of surgery to 24 hours after surgery complete (average surgical duration 2.5 hours).
  Cumulative 24-hr postoperative opioid consumption
Pain scores for the 1st 24 hours after surgery (Numeric Rating Scale Pain) | 1st 24 hours after completion of surgery.
  Numeric Rating Scale Pain prior to hospital discharge, 1 hour after arriving home, 4 hours after arriving home, 1 hour prior to going to sleep, 1 hour after waking up the next morning, 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Francis Salinas, MD, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States